CLINICAL TRIAL: NCT02190656
Title: Anterior Resection Syndrome Following Sphincter-preserving Surgery
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Other Study IDs: 009515
Record Dates: First submitted 2014-03-12; First posted 2014-07-15 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Anterior Resection Syndrome; Functional outcomes
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anterior resection: Patients having had an anterior resection for rectal cancer who are more than 12 months post surgery

SUMMARY:
Bowel cancer is the third most common cancer in the UK in both males and females. The rectum is the most commonly affected part of the bowel. Improvements in surgery have meant that many patients with rectal cancer can now undergo surgery that removes the rectum and avoids a permanent stoma. The operation that most patients have is an anterior resection of the rectum.

Unfortunately this surgery frequently leads to a change in bowel function, with patients suffering from incontinence, urgency and unpredictability a problem known as anterior resection syndrome. These problems are believed to be fairly common following surgery but follow up appointments have traditionally concentrated on ensuring that the cancer has not returned and have not reviewed functional outcomes in enough detail. Because of this we are unsure exactly how common the problems described are.

The proposed study will allow us to determine how many patients have ongoing symptoms following their surgery for rectal cancer. It will also allow us to use a newly developed scoring system the Low Anterior Resection Syndrome (LARS) score for the first time in a UK population, to ensure that it can accurately be used in the future to measure the problem and aid development of new therapies. An appreciation of the impact of symptoms on postoperative quality of life will encourage routine assessment of functional outcomes in clinical practice, allowing identification of patients who may benefit from treatment.

DETAILED DESCRIPTION:
One of the main aims when carrying out surgery for rectal cancer is to avoid patients ending up with a permanent stoma. The current standard operation for resection of the rectum is an anterior resection. A large proportion of the patients undergoing this procedure develop anterior resection syndrome, with significant alteration of their bowel habit, including urgency, incontinence and unpredictability. Many definitions for this problem have been used and until recently there was no specifically designed tool for measuring it. There has never been a large scale study in the UK to tell us how common the problem is. A meta-analysis combining results from small studies show marked variation in the frequency of symptoms ranging from 285%, mainly because of the different methods of assessment used in the studies.

The LARS score was recently developed by a research group in Denmark. Their results show that 45.9% of patients had major LARS at 12 months following surgery. This is nearly half of all patients in their sample and clearly represents an important problem.

Anterior resection syndrome is known to have a negative effect on quality of life. It is a multifactorial condition and is increased in patients have chemotherapy and radiotherapy. There are treatments available and also in development which may help patients. However in clinical practice, patients are not routinely asked about their functional outcome and the effect that these symptoms can have on patients' lives is often not discussed. The urgent need for further research into the longterm functional effects of treatments for cancer has been acknowledged by the National Institute for Health and Care Excellence (NICE) and the National Cancer Survivorship Initiative.

Determining baseline prevalence in the UK and validating the LARS score will allow accurate preoperative counselling of patients about functional outcomes following surgery for rectal cancer. It will facilitate comparison between populations, further helping to determine risk factors and aiding in development of therapeutic interventions. An appreciation of the impact of anterior resection syndrome on postoperative quality of life will encourage routine assessment of functional outcomes in clinical practice, allowing identification of patients who may benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having had an anterior resection for rectal cancer who are more than 12 months post surgery
* Patients who are more than 12 months post reversal of any defunctioning stoma
* Aged over 18 years

Exclusion Criteria:

* Any inclusion criteria not met
* Presence of a stoma
* Local recurrence of cancer
* Current adjuvant therapy
* Further rectal surgery after the initial operation
* Insufficient written English to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had an anterior resection for rectal cancer who are more than 12 months post surgery
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with no LARS; minor LARS and major LARS | At the time of questionnaire completion
  This will allow us to determine the prevalence of Low Anterior Resection Syndrome

SECONDARY OUTCOMES:
Correlation between LARS score and EORTC QLQ-C30 questionnaire score | At the time of questionnaire completion
  The association between the LARS score and The European Organization for Research and Treatment of Cancer (EORTC) generic quality of life questionnaire QLQC30 will be used to establish validity of the LARS score. Ability of the score to differ between patient groups known to differ in postoperative function (for example, those who have had radiotherapy and those who have not) will also be used to assess validity.

OTHER OUTCOMES:
LARS score in different age groups | At time of questionnaire completion
LARS score in participants who have had laparoscopic surgery and participants who have had open surgery | At time of questionnaire completion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Thaha, PhD FRCS, Study Chair — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom